CLINICAL TRIAL: NCT03132974
Title: Evaluation of Efficacy and Safety of Single and Multiple Therapy of Herbal Medicine/Chuna Therapy on Non-specific Chronic Low Back Pain: A Study Protocol for Multicenter, 3-arm, Randomized, Single Blinded, Parallel Group, Incomplete Factorial Design, Pilot Study -
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: Daejeon University (Other); Semyung University Korean Medicine Hospital in Chungju (Unknown); Woosuk University Oriental Medical Center (Unknown)
Responsible Party: Principal Investigator, Yun-Kyung Song, PhD, Gachon University Gil Oriental Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISEE_2017_LBP
Record Dates: First submitted 2017-04-19; First posted 2017-04-28 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SGHH (Experimental): Admission to Sogyeonghwalhyeol-tang granule
  Interventions: Drug: Sogyeonghwalhyeol-tang granule
- SGHH with manipulation therapy (Experimental): Admission to Sogyeonghwalhyeol-tang granule and manipulation therapy
  Interventions: Other: Sogyeonghwalhyeol-tang granule with manipulation procedure
- Placebo with manipulation therapy (Placebo Comparator)
  Interventions: Other: Placebo with manipulation procedure

INTERVENTIONS:
Drug: Sogyeonghwalhyeol-tang granule — Sogyeonghwalhyeol-tang herbal extract granule
  Arms: SGHH
Other: Sogyeonghwalhyeol-tang granule with manipulation procedure — Sogyeonghwalhyeol-tang herbal extract granule with manipulation procedure
  Arms: SGHH with manipulation therapy
Other: Placebo with manipulation procedure — Placebo granule with manipulation procedure
  Arms: Placebo with manipulation therapy

SUMMARY:
The Purpose of this trial is to investigate the efficacy and safety of herbal medicine with manipulation therapy on Korean Patients with Chronic Low Back Pain

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with chief complaint of low back pain in oriental rehabilitation medical center
* Age 19 - 65
* Patients who have 4 ~7 cm of VAS pain score;
* Ability to have normal communication
* Ability to give informed consent

Exclusion Criteria:

* Patients with pain duration of 3 months or less
* Patients with progressive neurologic deficit or severe neurologic symptoms by SLR test
* Patients diagnosed with serious pathology(s) which may cause low back pain (e.g. spinal metastasis of tumor(s), acute fracture, etc)
* Patients with spondylolisthesis or spondylolysis(diagnosed with grade II or higher level)
* Patients currently taking steroids, immunosuppressants, medicine for mental illness or other medication(s) that may interfere with study results
* Patients with history of spinal surgery
* Patients with more severe pain than pain caused by low back pain
* Those who do not (cannot) abide by treatment and follow up due to the mental illness such as behavior disorder, depression, anxiety neurosis etc.
* Patients with history of Medical Malpractice Case
* Patients with treatment history of low back pain within 1 month either KM or WM
* Patients participating in other clinical studies within 3 months
* Pregnant patients or patients with plans of pregnancy or lactating patients
* Patients disagree to sign the informed consent form
* Patients deemed unsuitable for participating the trial by the researchers

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Numeric Rating Scale of Pain | Screening Visit, At baseline, week 2, 4, 6, 8
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) assesses the patients' current level of pain.

SECONDARY OUTCOMES:
Change from Baseline in 'Roland Morris Disability Questionnaire' | Screening Visit, At baseline, week 2, 4, 6, 8
  This is a self-reported questionnaire consisting of 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, bending over, sitting, lying down, dressing, sleeping, self-care and daily activities.
Change from Baseline in European Quality of life 5 Dimension | Screening Visit, At baseline, week 2, 4, 6, 8
  The EQ-5D is an international, standardized, generic instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state.

OTHER OUTCOMES:
Change from baseline in pelvic incidence | At baseline, week 4, 8
  angle between the line perpendicular to the sacral plate and the line connecting the midpoint of the sacral plate to the bicoxofemoral axis.
Change from baseline in iliac crest height | At baseline, week 4, 8
  A measure of the vertical distance from the top of the iliac crest to the floor while the subject stands.
Change from baseline in lumbar gravity line | At baseline, week 4, 8
  created by first locating center of the L3 body & then droping a line downward from there, perpendicular to the bottom of the film.
Change from baseline in lumbar lordotic angle | At baseline, week 4, 8
  the angle between the top (superior surface) of the second lumbar vertebra and the bottom (inferior surface) of the fifth lumbar vertebra

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Kyung Song, PhD, Principal Investigator — Gachon University Gil Oriental Medical Hospital
Locations (1):
- Gachon University Gil Oriental Medicine Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko Y, Jang BH, Oh MS, Kim SJ, Ko YS, Ha IH, Lee EJ, Kim MR, Song YK, Ko SG. Evaluation of efficacy and safety of single and multiple therapy of herbal medicine/Chuna therapy on non-specific chronic low back pain: A study protocol for multicenter, 3-arm, randomized, single blinded, parallel group, incomplete factorial design, pilot study. Medicine (Baltimore). 2020 Jul 24;99(30):e21260. doi: 10.1097/MD.0000000000021260. PMID 32791704